CLINICAL TRIAL: NCT05208814
Title: A Parallel, Open, Single-dose Administration Phase I Study to Evaluate the Pharmacokinetics and Safety of TPN171H Tablets in Patients with Renal Insufficiency and Healthy Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety of TPN171H Tablets in Patients with Renal Insufficiency and Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Collaborators: Shanghai Institute of Materia Medica, Chinese Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPN171H-10
Record Dates: First submitted 2021-12-29; First posted 2022-01-26 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2023-02

CONDITIONS: Pulmonary Arterial Hypertension; Erectile Dysfunction
Keywords: TPN171H; renal insufficiency; Pharmacokinetics
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Erectile Dysfunction; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Renal Insuffiency (Experimental): Subjects with various degrees of renal insuffiency
  Interventions: Drug: TPN171H single dose
- healthy subjects (Experimental): healthy subjects
  Interventions: Drug: TPN171H single dose

INTERVENTIONS:
Drug: TPN171H single dose — 10 mg TPN171H taken once

SUMMARY:
To evaluate the effect of renal insufficiency on the pharmacokinetics of TPN171H tablets after single dose oral administration, so as to provide basis for formulating clinical medication plan for patients with renal insufficiency; To evaluate the safety of TPN171H tablets in patients with renal insufficiency and healthy subjects

DETAILED DESCRIPTION:
The study design of two centers, parallel, open and single dose administration is adopted. The experiment is carried out in two stages, whether or not to start the second stage is according to the test results of the first stage.

The first stage: there are two groups: severe renal insufficiency group and healthy subjects group. 8 subjects in each group (both male and female), a total of 16 cases.

The second stage: part A or part B. Part A: there are two groups: non dialysis end-stage renal disease (ESRD) group, with 8 subjects (both men and women), in the group with healthy subjects , there are 0-8 subjects.

Part B: there are three groups: mild renal insufficiency, moderate renal insufficiency and healthy subjects. There are 8 subjects (both male and female) in both mild renal insufficiency group and moderate renal insufficiency group, and 0-8 subjects (both male and female) in the healthy subjects group.

The initiation criteria of second stage study are: if auc0-t of subjects with severe renal insufficiency in the first stage is less than twice that of subjects with healthy subjects, And expected in the end of nephropathy If there is no significant increase in safety risk among (non dialysis) subjects, it is decided to start the second stage part A study instead of the second stage part B study according to the results of the first stage; if the auc0-t of subjects with severe renal insufficiency in the first stage is more than twice that of subjects with healthy subjects, it is decided whether to start the second stage part B study instead of the second stage part A study according to the results of the first stage.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old, both male and female;
2. Weight: male ≥ 50 kg, female ≥ 45 kg, 18 kg/m2 ≤ BMI ≤ 30 kg/m2 ;
3. Healthy subjects meet: GFR ≥ 90ml / min and < 130ml / min; the GFR of the subjects in the corresponding group meet the criteria of MDRD in the stage of renal function. Mild renal insufficiency (CKD 2 stage) : GFR : 60-89 mL/min; moderate renal insufficiency (CKD 3 stage) : GFR : 30-59mL/min; Severe renal insufficiency (CKD 4): GFR: 15-29 mL/min; renal failure (CKD 5) : GFR<15 mL/min；
4. Be able to understand the procedures and methods of this study, be willing to strictly abide by the clinical trial scheme, complete this trial, and voluntarily sign the informed consent.

Exclusion Criteria:

* Common exclusion criteria of each group:

  1. Dysphagia;
  2. Arrhythmia with clinical significance, or QTCF > 450ms (male) and QTCF > 470ms (female);
  3. Subjects with acute hepatitis, chronic liver disease, positive treponema pallidum antibody, positive HBV surface antigen, positive HCV antibody and positive HIV antibody; Or either ALT or AST is greater than 2 times the upper limit of the normal value, and the total bilirubin is greater than 1.5 times the upper limit of the normal value.
  4. Subjects with history of drug allergy, allergic constitution and family history of allergy;
  5. Subjects who have used drugs that affect the function of liver metabolic enzymes within 30 days before the start of the test, or those who need to use other drugs that may affect the absorption, distribution, metabolism and excretion of the tested drugs during the test;
  6. Subjects who drink too much (more than 8 cups a day, 1 cup = 250mL) of tea, coffee or caffeinated beverages within 6 months before screening; or those who consumed any food or beverage rich in caffeine and / or xanthine within 48 hours before the first administration of the study to the end of the test.
  7. Subjects who have a history of alcohol, tobacco and drug abuse; subjects whose alcohol breath test is positive, and urine drugs (morphine, tetrahydrocannabinol acid, methamphetamine, dimethylbisoxyamphetamine, ketamine) screening results are positive;
  8. Subjects who participated in the drug clinical trial within 3 months before the trial;
  9. Subjects who participate in blood donation within 3 months from the beginning of the test and the blood donation volume is ≥ 400mL or receive blood transfusion;
  10. Subjects who have undergone surgery within 4 weeks before screening, or plan to perform surgery during the study or within 2 weeks after the end of the study;
  11. Subjects who cannot tolerate venipuncture, or have a history of needle fainting and blood fainting;
  12. Women of childbearing age with positive pregnancy test, or pregnant and lactating women and subjects who are unwilling or unable to take physical contraceptives during the test;
  13. The researchers believe that subjects with any factors that are not suitable to participate in this trial.
* Exclusion criteria for healthy subjects:

  1. Subjects whose physical examination, vital signs, blood routine, blood biochemistry, urine routine, coagulation function, full chest positive film and 12 lead ECG, at least one of which is judged by the researcher to be abnormal and of clinical significance;
  2. Subjects whose systolic blood pressure < 85mmHg or > 140mmHg, diastolic blood pressure < 55mmHg or > 90mmHg;
  3. Subjects who have previous or existing diseases of liver, kidney, endocrine, digestive system, urinary system, cardiovascular system, nervous system, respiratory system (such as asthma, chronic obstructive bronchitis, etc.), blood and lymphatic system, nervous system (such as multiple headache), mental diseases and other diseases with clinical significance judged by the research doctor;
  4. Subjects who have used any drugs (including prescription drugs, over-the-counter drugs, vitamin supplements or Chinese herbal medicine) and health products within 2 weeks before screening;
* Exclusion criteria for subjects with renal insufficiency:

  1. 1 years before the start of the trial, subjects who have serious diseases such as cardiovascular, neuropsychiatric, digestive, respiratory, endocrine and other systems besides renal insufficiency basic diseases and their complications (such as diabetic nephropathy, renal anemia, renal hypertension, etc.).
  2. Subjects who have significant laboratory abnormalities related to renal insufficiency and its complications, which are clinically significant according to the judgment of the researcher;
  3. Subjects with diabetic nephropathy have a HbAlc > 8.5% and fasting blood glucose > 11.1mmol/L at least 4 weeks before treatment.
  4. The researcher believes that the subject's condition (such as blood pressure) is not suitable for the selection of this researcher;
  5. Subjects with renal insufficiency have no evidence of a history of chronic diseases lasting more than 1 months, including but not limited to chronic glomerulonephritis, benign glomerular arteriosclerosis, obstructive nephropathy or diabetes, and the results of the study indicate that the GFR of subjects may change significantly during the study period.
  6. During the period from 1 month before taking the test drug to the end of the study, the investigator judge that there is no stable scheme for the treatment of renal function insufficiency and its complications (medication type, dose or medication frequency, etc.);
  7. Subjects who have renal insufficiency with renal anemia, Hb < 80 g / L;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) | 72 hours or 120 hours after dosing
  Area under the curve (AUC) for plasma and urine following a single dose of TPN171H in subjects with renal insuffiency and healthy subjects.
Time to maximum plasma concentration (Tmax) | 72 hours or 120 hours after dosing
  Time to maximum plasma concentration (Tmax) for plasma and urine following a single dose of TPN171H in subjects with renal insuffiency and healthy subjects.
Maximum plasma concentration (Cmax) | 72 hours or 120 hours after dosing
  Maximum plasma concentration (Cmax) for plasma and urine following a single dose of TPN171H in subjects with renal insuffiency and healthy subjects.
Terminal half-life (t 1/2) | 72 hours or 120 hours
  Terminal half-life (t 1/2) for plasma and urine following a single dose of TPN171H in subjects with renal insuffiency and healthy subjects.
Apparent distribution volume (Vd) | 72 hours or 120 hours after dosing
  Apparent distribution volume (Vd) for plasma and urine following a single dose of TPN171H in subjects with renal mpairment and healthy subjects.
Clearance rate (CL) | 72 hours or 120 hours after dosing
  Clearance rate (CL) for plasma and urine following a single dose of TPN171H in subjects with renal insuffiency and healthy subjects.
Oral bioavailability (F) | 72 hours or 120 hours after dosing
  Oral bioavailability (F) for plasma and urine following a single dose of TPN171H in subjects with renal insuffiency and healthy subjects.
Adverse events | From administration of study drug through 8 days after administration of study drug
  Number of Participants With treatment-related Adverse Events and Serious Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Miao, Principal Investigator — West China Hospital; Ping Fu, Principal Investigator — West China Hospital; Xiaolan Yong, Principal Investigator — Chengdu Xinhua Hospital
Locations (2):
- China (2):
  - West China Hospital, Chengdu, Sichuan
  - Chengdu Xinhua Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No